CLINICAL TRIAL: NCT06700694
Title: The Effect of Technology-Assisted Early Mobilization Program Among Patients in the Intensive Care Units: a Randomized Controlled Trial
Brief Title: Technology-Assisted Early Mobilization Program Among Patients in the Intensive Care Units
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hsiao-Yean Chiu (Other)
Collaborators: Taipei Medical University Hospital (Other); National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor-Investigator, Hsiao-Yean Chiu, Professor, Taipei Medical University
Organization: Taipei Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202403085
Record Dates: First submitted 2024-11-01; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Intensive Care Unit Acquired Weakness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Technology-assisted early mobilization group (Experimental): Participants in the technology-assisted early mobilization group will receive protocol-oriented early mobilization program and technology-assisted, family-engaged in-bed activities within 72 hours of ventilator use.
  Interventions: Other: Technology-assisted, family-engaged in-bed activities; Other: Protocol-oriented early mobilization program
- Systematic early mobilization group (Active Comparator): Participants allocated to the systematic early mobilization group will receive the same protocol-oriented early mobilization program within 72 hours of ventilator use.
  Interventions: Other: Protocol-oriented early mobilization program
- Usual care group (No Intervention): Participants in the usual care group will receive routine rehabilitation treatment.

INTERVENTIONS:
Other: Technology-assisted, family-engaged in-bed activities — Technology-assisted, family-engaged in-bed activities include handgrip interactive games, virtual reality butterfly catching, virtual reality magic cube games, and immersive in-bed cycling, performed 20 minutes per session, twice daily, five days a week, primarily assisted by family members.
  Arms: Technology-assisted early mobilization group
Other: Protocol-oriented early mobilization program — The protocol-oriented early mobilization program is implemented based on the patient's muscle strength and the Intensive care unit Mobility Scale (IMS), including lying, sitting, standing, stepping, and walking, once daily for 20-60 minutes, five days a week, carried out by physiotherapist and researcher.
  Arms: Systematic early mobilization group; Technology-assisted early mobilization group

SUMMARY:
This single-blind, three-group parallel randomized controlled trial will involve 138 patients with critical illness, randomly assigned at a 1:1:1 ratio to the technology-assisted early mobilization group (46 patients), the systematic early mobilization group (46 patients), or the control group (46 patients). The technology-assisted early mobilization group will receive interventions within 72 hours of ventilator use. The interventions include protocol-oriented early mobilization program carried out by physiotherapist and researcher and technology-assisted in-bed activities primarily assisted by family members. The systematic early mobilization group will receive only the similar protocol-oriented early mobilization program within 72 hours of ventilator use. The control group will receive routine rehabilitation as usual. The primary outcomes include occurrence of intensive care unit-acquired weakness (ICUAW). Secondary outcomes include muscle strength, delirium, sleep status, clinical outcomes, activities of daily living, and quality of life. Measurements will be assessed on the day of enrollment, during the ICU stay, on the day of ICU discharge (or up to 28 days), on the day of hospital discharge, and six months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Being mechanically ventilated ≥ 24 hours
* Richmond Agitation-Sedation Scale (RASS): 0 to -1
* No vision, hearing, or body movements restriction
* With clear consciousness and ability to communicate in Chinese
* Expected to stay in the ICU > 96 hours.

Exclusion Criteria:

* Being pregnant, menopausal, or having a night shift within one month before admission to the ICU
* Have developed delirium before enrollment (ICDSC > 4)
* With acute physiology and chronic health evaluation (APACHE II) score > 25 after ICU admission within 24 hours
* With muscle weakness caused by severe acute brain injury (e.g., traumatic brain injury or stroke), spinal coral injury, other neuromuscular conduction diseases, or long-term bedridden or hemiplegia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of intensive care unit-acquired weakness (ICUAW) | On the day of enrollment and ICU discharge (or up to 28 days after enrollment).
  The occurrence of ICUAW will primarily be assessed using the Medical Research Council (MRC) scale. An MRC sum score of less than 48 indicates the presence of ICUAW.

SECONDARY OUTCOMES:
Muscle power | On the day of enrollment and ICU discharge (or up to 28 days after enrollment).
  Muscle power will be evaluated using the MRC scale, which assesses the strength of six bilateral muscle groups rated from 0 (complete paralysis) to 5 (normal strength) for each group. The total score ranges from 0 to 60.
Hand-grip strength | On the day of enrollment and ICU discharge (or up to 28 days after enrollment).
  Hand-grip strength will be measured using a hydraulic hand dynamometer. A strength of less than 11 kg for males and less than 7 kg for females indicates the presence of ICUAW. This outcome will be used to assess the occurrence of ICUAW, as determined by the MRC sum score, concurrently.
Delirium | Through intervention completion, up to 28 days.
  Delirium is assessed by the Intensive Care Delirium Screening Checklist (ICDSC), which includes eight items. Each item is scored as absent (0) or present (1), with total score ranging from 0 to 8. A score of ≥ 4 indicates the presence of delirium. The scoring is based on observations during every nursing shift.
Subjective sleep status | Through intervention completion, up to 28 days.
  Richards-Campbell Sleep Questionnaire (RCSQ) will be used to assess subjective sleep quality on a visual analog scale among patients in the ICU. The total score is calculated with a formula and categorized into four levels: < 26 is very poor, 26-50 is poor, 51-75 is good, and > 76 is excellent.
Objective sleep status | Through intervention completion, up to 28 days.
  Objective sleep status will be evaluated by SOMNOwatch™, which can extract not only sleep related parameters but also calculate sleep stages using additional electroencephalography (EEG) sensors.
Functional Status | On the day of enrollment and ICU discharge (or up to 28 days after enrollment).
  Functional Status Score for the Intensive Care Unit (FSS-ICU) is used to assess the functional status of patients in the ICU. Patient's performance of five functional movements will be rated from 0 to 7. The total score ranges from 0 to 35, with higher scores indicating better functional status.
Duration of ventilation use | On the day of hospital discharge (expected up to 3 month).
  The duration of ventilation use is specified the accumulated days of using mechanical ventilation with endotracheal tube in the ICU for this hospitalization. This outcome will be recorded from the hospital's electronic system.
Length of stay in the ICU | On the day of hospital discharge (expected up to 3 month).
  The length of stay in the ICU will be recorded from the hospital's electronic system.
Length of stay in the hospital | On the day of hospital discharge (expected up to 3 month).
  The total length of stay in the hospital will be recorded from the hospital's electronic system.
Adverse event | Through intervention completion, up to 28 days.
  Any adverse events occur during the intervention session.
Activities of daily living (ADL) | On the day of ICU discharge (up to 28 days after enrollment), hospital discharge (expected up to 3 month), and six-month after hospital discharge.
  The ADL will be assessed by the Barthel Index. The total score ranges from 0 to 100. A score of ≥ 70 indicates independent daily living abilities.
Sleep quality | On the day of hospital discharge (expected up to 3 month) and six-month after hospital discharge.
  The Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep quality over the past month. Score ranges from 0 to 21, with a score > 5 indicating poor sleep quality; higher scores reflect worse sleep quality.
Quality of life (QoL) | On the day of hospital discharge (expected up to 3 month) and six-month after hospital discharge.
  The EuroQol Five-Dimensional Five-Level Scale (EQ-5D-5L) is used to evaluate health-related QoL. The health status classification comprises five dimensions, each with five levels, calculated using specific values. The vertical analog scale assesses the patient's overall evaluation of their current health status, ranging from 0 to 100. Higher scores indicate greater QoL.